CLINICAL TRIAL: NCT01938274
Title: Establishing Appropriate Activity Expectations After Total Joint Replacement
Brief Title: Leisure Expectations About Physical Activity Study
Acronym: LEAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment never started
Sponsor: West Virginia University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dina L Jones, PT, PhD, Professor, West Virginia University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: R24HS018622 (AHRQ)
Record Dates: First submitted 2013-02-12; First posted 2013-09-10 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
Keywords: Hip; Knee; Osteoarthritis; Arthroplasty; Physical Activity; Expectations; Leisure Activity
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Osteoarthritis; Motor Activity | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational intervention (Experimental): Patients in this group will receive a brief educational intervention to assist them in setting the appropriate expectations for leisure activity after surgery with respect to the type, amount, intensity, and duration of activity.
  Interventions: Other: Educational intervention
- Control group (No Intervention): No intervention will be received. Patients will receive a written version of the education intervention at the end of the study.

INTERVENTIONS:
Other: Educational intervention — A 30-minute discussion and slide presentation with a trained member of the research team.
  Arms: Educational intervention

SUMMARY:
To pilot test an activity-focused intervention that educates patients undergoing total hip (THA) or total knee (TKA) arthroplasty due to osteoarthritis about the appropriate type, frequency, intensity, and duration of expected leisure activities after surgery and to determine if the intervention changed expectations.

DETAILED DESCRIPTION:
Consecutive patients, aged 45 years and older, who are scheduled for primary total hip or knee arthroplasty due to osteoarthritis will be randomized to an intervention or control (no intervention) group. All patients will be interviewed by telephone prior to the intervention, by an interviewer blinded to group status, to collect data on current leisure activity and expected activity at 6 months after surgery. Patients will also complete a questionnaire to collect data on sociodemographic characteristics, comorbidities (American Academy of Orthopaedic Surgeons Comorbidity Index), pain intensity (0-10 scale), health-related quality of life (SF-12), hip-/knee-specific outcomes (Hip Dysfunction and Osteoarthritis Outcome Score/Knee Injury and Osteoarthritis Outcome Score), general expectations (Hospital for Special Surgery Total Hip/Knee Replacement Expectations Surveys), and stage of readiness for change.

All patients will receive usual medical care before surgery and visit the clinic to meet with the surgeon and nurse/physician assistant, and undergo pre-operative laboratory testing. Patients in the intervention group will also meet with a member of the research team to complete a 10-item pre-test, to assess knowledge of the key concepts in the intervention, and then be presented with a 20-minute slide presentation. The presentation will educate patients on the: 1) definition of physical activity and its associated health benefits for the general population and people with arthritis, (2) 2008 Physical Activity Guidelines for Americans, 3) appropriate types of aerobic activities that patients should engage in after THA/TKA (e.g., no- or low-impact activities), (4) appropriate intensity level for activities after THA/TKA (e.g., at least moderate intensity), (5) appropriate duration of participation in activities (e.g., in increments of 10 or more minutes), and (6) the appropriate amount of activity per week (e.g., ≥ 2.5 hours [150 minutes]).

Patients will then complete a satisfaction survey that will provide feedback on the content, format, and length of the intervention, and a post-test to measure mastery of the intervention material. The post-test will contain the same questions as the pre-test, but in a different order. The control group will not meet with the research team during their pre-operative visit. The control group will receive a written version of the intervention at the end of the study.

All patients will be re-interviewed by telephone one week after their visit to reassess leisure activity expectations. Data analyses will be conducted to determine: 1) the direction and magnitude of change expected in leisure activity between baseline and 6 months, 2) the change in the proportion of patients who expect to meet national physical activity guidelines 6 month after surgery, and 3) whether or not the intervention modified the type, frequency, duration, or intensity of expected leisure activity from pre- to post-administration.

ELIGIBILITY:
Inclusion Criteria:

* The study includes male or female patients, aged 45 years and older who are scheduled for primary total hip or knee arthroplasty due to osteoarthritis.

Exclusion Criteria:

* Patients will be excluded from the study if the surgery is being performed for diagnosis other than osteoarthritis.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Change in type, frequency, intensity, and duration of expected leisure activities from pre- to post-intervention. | One-week prior to the educational intervention (Pre) (approximately 3-4 weeks before surgery) and one-week after the educational intervention (Post) (approximately 1-2 weeks before surgery).
  The Historical Leisure Activity Questionnaire will be used to measure expected physical activity before and after the intervention

SECONDARY OUTCOMES:
Change in the proportion of patients who expect to meet nationally recommended physical activity levels 6 months after surgery. | One-week prior to the educational intervention (Pre) (approximately 3-4 weeks before surgery) and one-week after the educational intervention (Post) (approximately 1-2 weeks before surgery).
  The Historical Leisure Activity Questionnaire will be used to determine if patients expect to meet the nationally recommended physical activity levels 6 months after surgery (i.e., 2.5 hours or more of at least moderate-intensity aerobic activity per week in bouts of 10 or more minutes).
Direction and magnitude of change expected in leisure activity between baseline (i.e., current activity) and 6 months | Baseline (approximately 3-4 weeks before surgery)
  Expected activity at 6 months - baseline activity = expected change in activity

CONTACTS AND LOCATIONS:
Overall Officials: Dina L. Jones, PT, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No